CLINICAL TRIAL: NCT04441827
Title: The Study Aims to Evaluate Effectiveness of Pranayama and Deep Breathing Exercise in Reducing Fatigue and Insomnia in Patients Receiving Radiotherapy Due to Breast Cancer.
Brief Title: Using Pranayama and Deep Breathing Exercises to Reduce Cancer-Related Fatigue and Insomnia During Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Fatma Gündoğdu, Principal İnvestigator, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UPDBERCRFIDR
Record Dates: First submitted 2020-06-12; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer; Fatigue; Insomnia
Keywords: Breast cancer; Fatigue; Insomnia; Pranayama; Radiotherapy; Breathing exercises
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Sleep Initiation and Maintenance Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Usual care
- Pranayama (Experimental): Pranayama breathing exercise
  Interventions: Other: breathing exercise
- Deep breathing exercise (Experimental): Deep breathing exercise
  Interventions: Other: breathing exercise

INTERVENTIONS:
Other: breathing exercise — Pranayama Group Breathing Exercises Step One:Focusing on breathing (1 minute) Step Two: Alternative nasal breathing (3 minutes) Step Three: Refreshing breath (3 minutes) Step Four: Humming bee breath (2 minutes) Step Five: Focusing on breathing (1 minute)
  Arms: Deep breathing exercise; Pranayama

SUMMARY:
The study aims to evaluate the effectiveness of pranayama and deep breathing exercise in reducing fatigue and insomnia in patients receiving radiotherapy due to breast cancer. The randomized controlled interventional study was carried out with 60 patients divided into the pranayama (20), deep breathing exercise (20) and control group (20). Data were collected with the Piper Fatigue Scale (PFS), the Pittsburgh Sleep Quality Index (PSQI) and the Visual Analog Scale (VAS).

DETAILED DESCRIPTION:
Study sample The study population consisted of patients diagnosed with breast cancer, who received radiotherapy in the radiation oncology unit of a hospital in Ankara, between June 01, 2017 and January 31, 2019.

At least three additional volunteers (16%) for each group were added, considering monitoring and data loss during the follow-up. Thus, the number of subjects was determined as 63 individuals (21 for each group).

Of the 63 patients, one wanted to interrupt the treatment and two did not want to continue in the study, hence the study was concluded with 20 patients in each group (60 patients).

Instruments Fatigue Visual Analog Scale (VAS) Score Piper Fatigue Scale (PFS) Insomnia Visual Analog Scale (VAS) Score Pittsburgh Sleep Quality Index (PSQI) Questionnaire on Patients' Opinions of the Exercises Patients in the pranayama, deep breathing exercise and control group were evaluated six times in terms of fatigue and insomnia VAS scores. PFS and PSQI were evaluated once prior to and after the 25-day session of radiotherapy treatment.

Interventions Protocols for pranayama and deep breathing exercises were prepared Pranayama and Deep Breathing Exercise Groups: The patients were taught pranayama and deep breathing exercises by the researcher before the radiotherapy started. The patients were observed performing these exercises for 10 minutes after each radiotherapy session (25 days) accompanied by the researcher in a quiet room within the radiotherapy unit containing two couches and a chair.

Control Group: The patients in this group did not receive any intervention.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18 years,
* who underwent breast resection or modified radical mastectomy,
* were planned for radiotherapy for the chest wall/breast and lymphatic area, had Stage II-III breast cancer according to the TNM (Tumor diameter, Node, Metastasis) classification system,
* had a hemoglobin (HgB) level of 10 gm/dL and above,
* scored 0 or 1 on the ECOG (Eastern Cooperative Oncology Group) Performance Scale
* who agreed to participate in the study were included in the sample.

Exclusion Criteria:

* having any problems that would prevent communication,
* having stage IV breast cancer according to the TNM classification system,
* using opioids or sedating drugs,
* scoring above 1 on the ECOG Performance Scale,
* having psychiatric illnesses,
* taking yoga/pranayama/deep breathing exercise lessons before or having done these exercises prior to diagnosis,
* having recurrent breast cancer
* being unable to perform the exercises due to physical inability/respiratory distress.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Fatigue Visual Analog Scale (VAS) Score | Before radiotherapy
  This scale which evaluates the severity of fatigue, was scored as follows: no fatigue= 0 points, mild fatigue= 1-3 points, moderate fatigue= 4-6 points, severe fatigue= 7-9 points and unbearable fatigue= 10 points.
Fatigue Visual Analog Scale (VAS) Score | First week
  This scale which evaluates the severity of fatigue, was scored as follows: no fatigue= 0 points, mild fatigue= 1-3 points, moderate fatigue= 4-6 points, severe fatigue= 7-9 points and unbearable fatigue= 10 points.
Fatigue Visual Analog Scale (VAS) Score | Second week
  This scale which evaluates the severity of fatigue, was scored as follows: no fatigue= 0 points, mild fatigue= 1-3 points, moderate fatigue= 4-6 points, severe fatigue= 7-9 points and unbearable fatigue= 10 points.
Fatigue Visual Analog Scale (VAS) Score | Third week
  This scale which evaluates the severity of fatigue, was scored as follows: no fatigue= 0 points, mild fatigue= 1-3 points, moderate fatigue= 4-6 points, severe fatigue= 7-9 points and unbearable fatigue= 10 points.
Fatigue Visual Analog Scale (VAS) Score | Fourth week
  This scale which evaluates the severity of fatigue, was scored as follows: no fatigue= 0 points, mild fatigue= 1-3 points, moderate fatigue= 4-6 points, severe fatigue= 7-9 points and unbearable fatigue= 10 points.
Fatigue Visual Analog Scale (VAS) Score | Fifth week
  This scale which evaluates the severity of fatigue, was scored as follows: no fatigue= 0 points, mild fatigue= 1-3 points, moderate fatigue= 4-6 points, severe fatigue= 7-9 points and unbearable fatigue= 10 points.
İnsomnia Visual Analog Scale (VAS) Score | Before radiotherapy
  The scoring system of this scale was as follows: no insomnia= 0 points, mild insomnia= 1-3 points, moderate insomnia= 4-6 points, severe insomnia= 7-9 points and unbearable insomnia= 10 points.
İnsomnia Visual Analog Scale (VAS) Score | First week
  The scoring system of this scale was as follows: no insomnia= 0 points, mild insomnia= 1-3 points, moderate insomnia= 4-6 points, severe insomnia= 7-9 points and unbearable insomnia= 10 points.
İnsomnia Visual Analog Scale (VAS) Score | Second week
  The scoring system of this scale was as follows: no insomnia= 0 points, mild insomnia= 1-3 points, moderate insomnia= 4-6 points, severe insomnia= 7-9 points and unbearable insomnia= 10 points.
İnsomnia Visual Analog Scale (VAS) Score | Third week
  The scoring system of this scale was as follows: no insomnia= 0 points, mild insomnia= 1-3 points, moderate insomnia= 4-6 points, severe insomnia= 7-9 points and unbearable insomnia= 10 points.
İnsomnia Visual Analog Scale (VAS) Score | Fourth week
  The scoring system of this scale was as follows: no insomnia= 0 points, mild insomnia= 1-3 points, moderate insomnia= 4-6 points, severe insomnia= 7-9 points and unbearable insomnia= 10 points.
İnsomnia Visual Analog Scale (VAS) Score | Fifth week
  The scoring system of this scale was as follows: no insomnia= 0 points, mild insomnia= 1-3 points, moderate insomnia= 4-6 points, severe insomnia= 7-9 points and unbearable insomnia= 10 points.
Piper Fatique Scale | Before radiotherapy
  Piper Fatique Scale scale consisted of 22 items and evaluated the patient's subjective fatigue perception with four subdimensions. Each item was scored between 0 and 10. A high score obtained from the scale indicated a high level of perceived fatigue.
Piper Fatique Scale | Fifth week
  Piper Fatique Scale consisted of 22 items and evaluated the patient's subjective fatigue perception with four subdimensions. Each item was scored between 0 and 10. A high score obtained from the scale indicated a high level of perceived fatigue.
Pittsburgh Sleep Quality Index | Before radiotherapy
  Pittsburgh Sleep Quality Index is a self-report-based screening and evaluation tool that provides detailed information on sleep quality and type and severity of sleep disorder in the past month.The total PSQI score could vary from 0 to 21. A PSQI score over 5 points indicated that the person suffered serious problems in at least two areas related to sleep or that they suffered mild to moderate problems in more than three areas
Pittsburgh Sleep Quality Index | Fifth week
  Pittsburgh Sleep Quality Index is a self-report-based screening and evaluation tool that provides detailed information on sleep quality and type and severity of sleep disorder in the past month.The total PSQI score could vary from 0 to 21. A PSQI score over 5 points indicated that the person suffered serious problems in at least two areas related to sleep or that they suffered mild to moderate problems in more than three areas

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yildirim Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Messer S, Oeser A, Wagner C, Wender A, Cryns N, Scherer RW, Mishra SI, Monsef I, Holtkamp U, Andreas M, Brockelmann PJ, Ernst M, Skoetz N. Yoga for fatigue in people with cancer. Cochrane Database Syst Rev. 2025 May 27;5(5):CD015520. doi: 10.1002/14651858.CD015520. PMID 40421669
- [Derived] Gundogdu F, Kocasli S. The Effects of Pranayama or Deep Breathing Exercises on Fatigue and Sleep Quality in Women Receiving Radiation Therapy for Breast Cancer. Oncol Nurs Forum. 2023 Jun 15;50(4):509-520. doi: 10.1188/23.ONF.509-520. PMID 37677752